CLINICAL TRIAL: NCT02200510
Title: Patient-Provider Interventions to Improve Transition to Adult Care in SCD
Brief Title: Patient-Provider Tools to Improve the Transition to Adult Care in Sickle Cell Disease
Acronym: iTransition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5K07HL108720 (NIH)
Record Dates: First submitted 2014-07-21; First posted 2014-07-25 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Sickle Cell Disease
Keywords: Anemia, Sickle Cell; Transition to Adult Care; Self Care; Personal Electronic Health Records; Adolescent; Young Adult; Disease Management; Physician-Patient Relations
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-Management Group (Other): Self-management intervention for Adolescents with SCD - 6 week self-management group
  Interventions: Behavioral: Self-management intervention for Adolescents with SCD
- Patient Portal (Other): Patient Portal Intervention for Adolescents with SCD - 6 week individual patient portal intervention
  Interventions: Behavioral: Patient Portal Intervention for Adolescents with SCD

INTERVENTIONS:
Behavioral: Self-management intervention for Adolescents with SCD — Chronic Disease Self-Management Program
  Arms: Self-Management Group
Behavioral: Patient Portal Intervention for Adolescents with SCD — MyChart for SCD intervention
  Arms: Patient Portal

SUMMARY:
The purpose of the study is to develop patient-provider clinical support tools to improve clinical practice, patient self-management, and disease outcomes in sickle cell disease during transition to adult care. The investigators hypothesize that these clinical support tools (patient tool, provider tool, and patient/parent web-based portal) will be feasible, user friendly, and beneficial. The investigators hypothesize that participants will demonstrate better disease self-efficacy at the end of the 6 week intervention and maintain these gains during the follow-up period (up to 1 year post-intervention).

DETAILED DESCRIPTION:
The purpose of the study is to develop patient-provider clinical support tools to improve clinical practice, patient self-management, and disease outcomes in sickle cell disease during transition to adult care.

ELIGIBILITY:
Inclusion Criteria:

* Have sickle cell disease (SCD)
* Between the ages of 13 and 24
* Receive care at Cincinnati Children's Hospital Medical Center, University Hospital, University of Cincinnati Med Peds Practice, a practice in the Ohio Valley SCD Network, or another local provider
* Parent/caregiver of a patient with SCD age 13-24 years

Exclusion Criteria:

* Below age 13
* Have significant health complication(s) that would interfere with completion of the intervention (by physician report)
* Have significant cognitive or developmental disabilities (by parent or physician report) due to high demand on participants to understand questions
* Are not a patient at Cincinnati Children's Hospital Medical Center, University Hospital, University of Cincinnati Med Peds Practice, a practice in the Ohio Valley SCD Network, or another local provider
* Are not a parent/caregiver of a patient with SCD age 13-24 years

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2011-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori E Crosby, PsyD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crosby LE, Smith T, Parr WD, Mitchell MJ. The Community Engagement and Translational Research Speaker Series: An Innovative Model of Health Education. J Community Med Health Educ. 2013 Jul 24;3:1000227. doi: 10.4172/2161-0711.1000227. PMID 25414800
- [Background] Edwards R, Telfair J, Cecil H, Lenoci J. Reliability and validity of a self-efficacy instrument specific to sickle cell disease. Behav Res Ther. 2000 Sep;38(9):951-63. doi: 10.1016/s0005-7967(99)00140-0. PMID 10957829
- [Result] Crosby LE, Joffe NE, Dunseath LA, Lee R. Design Joins the Battle Against Sickle-cell Disease. Des Manage Rev. 2013 Summer;24(2):48-53. doi: 10.1111/drev.10241. No abstract available. PMID 25414599
- [Result] Crosby, L.E., Hudepohl, M., Kalinyak, K., Britto, M., Goldstein, A., Brown, K., Culp, A., & Joiner, C. H. (2013). Impact of use of a disease-specific patient portal on transition readiness and quality of life in adolescents with sickle cell disease [Abstract]. Blood, 122(21), 2982.
- [Result] Crosby, L. E., Joffe, N., Kalinyak, K., Bruck, A. & Joiner, C. H. (2013). Six-month data from a pilot self-management intervention for adolescents with sickle cell disease [Abstract]. Blood, 122(21), 1675.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Self-Management Group | Patient Portal
Started | 31 (Number who only completed self-management or completed it before portal (could do 6 months later).) | 47 (Number who only completed portal or completed it before self-management (could do 6 months later).)
Completed | 22 (This is the number of participants with baseline and post data.) | 44 (This number is the number of participants with both baseline and post data.)
Not Completed | 9 | 3
Not completed — Death | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 7 | 1
Not completed — potential COI - joined study team | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed baseline measures
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-Management Group | Patient Portal | Total
Number analyzed (Participants) | 22 | 44 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 26 | 39
  Between 18 and 65 years | 9 | 18 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.77 (2.22) | 18.82 (2.72) | 18.795 (2.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 24 | 34
  Male | 12 | 20 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 44 | 66
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 44 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on Disease Self-efficacy Measure at 6 Weeks
Description: Name of Measure: Sickle Cell Self-Efficacy Scale (SCSES). Construct: sickle cell self-efficacy (disease specific self-efficacy) 9 item measure of sickle cell disease self-efficacy (likert scale from 1 [not at all sure] to 5 [very sure]) developed by Edwards (see References).
  Responses on items are summed to compute a total score. Minimum score: 9 Maximum score: 45 Higher scores represent higher sickle cell self-efficacy (better outcome).
Time Frame: baseline, 6 weeks (post-intervention)
Population: Participants with completed baseline and post measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-Management Group | Patient Portal
Number analyzed (Participants) | 22 | 44
units on a scale | 33.2 (5.49) | 33.09 (7.10)
Statistical Analysis 1: Comparison: Self-Management Group; Test type: Equivalence — Because this was a pilot study, the goal was to detect effects sizes for a larger R01 or R21; p = 0.575, ANOVA; Mean Difference (Final Values) = 0.33
Statistical Analysis 2: Comparison: Patient Portal; Test type: Equivalence — Because this was a pilot study, the goal was to detect effects sizes for a larger R01 or R21; p = 0.721, ANOVA; Mean Difference (Final Values) = .138

ADVERSE EVENTS:
Time Frame: During the 6 months participants were enrolled in the study.
Description: An adverse event (AE) for the current study is an unfavorable medical occurrence in a participant temporally associated with the subject's participation in the research, whether or not considered related to the subject's participation in the research. A serious adverse event (SAE) may or may not result in death, be life threatening, or require hospitalization. Since this population has frequent hospitalizations, only unexpected adverse events were reported here.
Arm/Group | Self-Management Group | Patient Portal
All-Cause Mortality (participants affected / at risk) | 1/22 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/44
Other Adverse Events (participants affected / at risk) | 0/22 | 0/44

LIMITATIONS AND CAVEATS:
Pilot feasibility studies with convenience samples.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No